CLINICAL TRIAL: NCT04780139
Title: Ultrasonographic Evaluation of Internal Jugular Vein Cross Sectional Area for Prediction of Post Spinal Hypotension in Patients Undergoing Orthopedic Surgeries
Brief Title: Ultrasonographic Evaluation of Internal Jugular Vein Cross Sectional Area for Prediction of Post Spinal Hypotension
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Walid Nofal, Assisstant professor, Ain Shams University
Other Study IDs: FMASU R 25/2020/2021
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Post-spinal Anesthesia Hypotension
Keywords: internal jugular vein; ultrasound; spinal anesthesia; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonographic Evaluation of Internal Jugular Vein Cross Sectional Area — Measuring the internal jugular vein cross section area and relate this to the incidence of hypotension after spinal anesthesia.

SUMMARY:
The aim of this study is to evaluate the efficacy of internal jugular cross sectional area for predicting the occurrence of PSAH.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of internal jugular cross sectional area for predicting the occurrence of PSAH. Spinal anaesthesia is frequently used in daily clinical practice. Postspinal anaesthesia hypotension (PSAH) is a common side effect with an incidence of 15.3 to 33% that may result in organ hypoperfusion and ischaemic events. Patients' susceptibility to intraoperative hypotension can be influenced by the sensory block level, age, preoperative volume status , physical status, pre-operative medications and fasting.

PSAH due to spinal blockade is principally a consequence of diminished systemic vascular resistance after blockade of preganglionic sympathetic fibres. Many attempts have been tried to prevent PSAH, such as intravenous volume preload or prophylactic vasopressors. However, fluid infusion has been proved to lower the incidence of PSAH and significantly decrease vasopressor requirements. At the same time, empirical volume loading carries the potential of volume overload, particularly in patients with cardiac disease. Consequently, the search for predictors of PSAH is becoming mandatory to avoid blind volume loading and reserve it only for patients who are expected to develop PSAH. .

.

ELIGIBILITY:
Inclusion Criteria:

* patients more than 40 years of age.
* American Society of Anesthesiologists' (ASA) physical status 1 or 2.
* scheduled for elective surgery under spinal anaesthesia in the supine position.

Exclusion Criteria:

* BMI more than 35 kg m2.
* taking angiotensin converting enzyme inhibitors.
* pregnant women.
* emergency cases.
* absolute or relative contraindications to spinal anaesthesia.
* Also, patients with a baseline arterial systolic blood pressure less than 90 mmHg or mean arterial blood pressure (MBP) less than 70 mmHg will be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients more than 40 years of age with American Society of Anesthesiologists' (ASA) physical status 1 or 2 who will be scheduled for elective orthopedic surgery under spinal anaesthesia in the supine position
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Predictive value of internal jugular vein (IJV) cross sectional area. | 30 minutes
  The primary outcome is to evaluate the predictive value of internal jugular diameter cross sectional area for detecting PSAH

CONTACTS AND LOCATIONS:
Overall Officials: Sanaa Farag Mahmoud, MD, Principal Investigator — Anesthesiology Department, Faculty of Medicine, Ain Shams University; Eman Sabek, MD, Principal Investigator — Radiology department, National Centre of Radiation Research and Technology, Atomic Energy Authority; WALID Nofal, MD, Principal Investigator — Anesthesiology department, Faculty of Medicine, Ain Shams Unive
Locations (1):
- Ain Shams University hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No